CLINICAL TRIAL: NCT05929898
Title: Bridging Scales to Understand Endogenous Neuromodulation and Its Regulation
Brief Title: MRI Neurofeedback and Brain Circuits Related to Motivation in Healthy Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00112672; 1R01MH131667-01 (NIH)
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-05

CONDITIONS: Motivation; Memory; Self-regulation
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intentional Versus Cue-Evoked Midbrain Activation (Experimental): Participants meeting study inclusion will be scheduled for two sessions: one baseline behavioral visit and an fMRI session to assess the ability to self-stimulate VTA activation. Session one will include a battery of cognitive assessments and a demonstration of the reward-based learning task in session two. The experimental imaging task session will be done within one week of session one. Participants will been randomly split into two group: group one will complete a reward-based learning task before the VTA activation task and group two will complete reward task after VTA activation. During the VTA activation task, participants will be instructed to achieve a heightened state of motivation using personally relevant thoughts and imagery.
  Interventions: Behavioral: Ventral tegmental area of dopaminergic midbrain (VTA) fMRI neurofeedback
- Intentional Midbrain Activation Effects on Effort-Based Decision Making (Experimental): Participants will be randomly assigned to an MRI group or a behavioral control group. All participants will complete an effort-based learning task and a series of questionnaires in session one. Session two may include an MRI based on group assignment. Participants in the MRI group will complete the VTA activation task. Following, they will complete the effort task and questionnaires a second time. The behavioral control group will complete a second session consisting of the effort task and questionnaires.
  Interventions: Behavioral: Ventral tegmental area of dopaminergic midbrain (VTA) fMRI neurofeedback
- Intentional Midbrain Activation Effects on Motivated Memory (Experimental): Participants will take part in four sessions: visit 1-baseline + memory encoding, visit 2-memory retrieval, visit 3-memory encoding, visit 4-memory retrieval). Encoding and retrieval of the memoranda will occur 24 hours apart. Study visits will take place no more than 7 days apart. One group of participants will complete all sessions at the Center for Cognitive Neuroscience. The remainder of participants will complete the encoding sessions in the MRI machine, .
  Interventions: Behavioral: Ventral tegmental area of dopaminergic midbrain (VTA) fMRI neurofeedback

INTERVENTIONS:
Behavioral: Ventral tegmental area of dopaminergic midbrain (VTA) fMRI neurofeedback — fMRI neurofeedback training of sustained midbrain/VTA activation via motivational imagery.

SUMMARY:
The purpose of this research study is to understand how healthy individuals self-regulate motivation by observing brain activity using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Neuromodulatory nuclei detect and transform brain network activity into simpler signals, then send neurotransmitters back out to large-scale brain networks to change their function. Such nuclei are centrally implicated in mental disorders and adaptive resilience, and their regulation remains an untapped resource for interventions. The purpose of this study is to understand how neuromodulatory nuclei detect and in turn influence distributed patterns of brain activity to impact behavior. In order to understand their regulation and effects on brain function, the investigative team has developed novel neuroimaging, behavioral, and analytic methods. These methods include: training participants to endogenously self-regulate dopaminergic midbrain and then relating midbrain activation to memory-conducive states, effort exertion, and decision making.

If the aims of this project are achieved, the investigators will have methods for regulating midbrain noninvasively, an improved understanding of its impact on learning and motivated behavior, and reliable cognitive strategies for a wide array of interventions across educational and clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Male or female
* Right-handed
* In good general health
* Women of childbearing capacity: use of effective method of birth control

Exclusion Criteria:

* Current or diagnosis within past six months of an DSM-V Axis I or Axis II disorder (self-reported)
* CES-D score of 20 or higher (indicating significant current depression symptoms)
* Current or past six month use of prescription medications indicated for psychiatric conditions (e.g.,depression, anxiety)
* Current serious medical illness (self-reported)
* Head injury resulting in loss of consciousness
* For participants age > 59 years, a total scaled score < 8 on the Dementia Rating Scale-2.
* A clinically-defined neurological disorder including, but not limited to:
* Any condition likely to be associated with increased intracranial pressure
* Space occupying brain lesion
* History of stroke
* Transient ischemic attack within two years
* Cerebral aneurysm
* Dementia
* Mini Mental Status Exam (MMSE) score of <24
* Parkinson's disease
* Huntington's disease
* Multiple sclerosis
* Presence of cochlear implants or other implanted electronic devices or non-removable metal (e.g., non-removable piercing, IUD)
* History of an eye injury involving metal. Participants who worked with metal may be allowed to participate on a case-by-case basis with prior written approval from BIAC.
* Claustrophobia or unwillingness to tolerate the confinement associated with being in the MRI scanner.
* Weight of more than 250 pounds

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Percent signal change in VTA BOLD activation | During the MRI scan, approximately 2 hours

SECONDARY OUTCOMES:
Change in effort-based decision making, as measured by the Effort Expenditure for Reward Task (EEfRT) | During the MRI scan, approximately 2 hours
  Decisions to exert effort.
Change in motivated memory, as measured by the Monetary Incentive Encoding task (MIE) | During the MRI scan, approximately 2 hours
  Improved motivated memory formation.

CONTACTS AND LOCATIONS:
Overall Officials: R. Alison Adock, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Center for Cognitive Neuroscience, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No